CLINICAL TRIAL: NCT04251221
Title: Measuring the Neuroimmune Response to Alcohol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Ansel Hillmer, Assistant Professor of Radiology and Biomedical Imaging and of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000024444; 1U54AA027989-01 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Drinkers (Experimental): Aim 1:
  A baseline PET scan with [11C]PBR28, a TSPO-specific radioligand, will be conducted with moderate drinkers. Next, subjects will drink a fixed alcohol dose, followed a post-alcohol [11C]PBR28 PET scan timed to capture acute neuroimmune response. [11C]PBR28 distribution volumes (VT), which are proportional to TSPO number, will be measured throughout the brain. We will test the hypothesis that acute alcohol robustly increases [11C]PBR28 VT, consistent with microglial activation. The percent change in [11C]PBR28 VT (ΔVT) from baseline will quantify the magnitude of neuroimmune response.
  Interventions: Drug: Oral Alcohol Challenge
- Alcohol Use Disorder (AUD) (Experimental): Aim 2:
  AUD subjects will participate in the study design described in Aim 1 (a baseline [11C]PBR28 PET scan, drink a fixed alcohol dose, followed by a post-alcohol [11C]PBR28 PET scans). The magnitude of neuroimmune response, quantified by ΔVT, will be compared between moderate drinkers and individuals with AUD to test the hypothesis that the neuroimmune response to alcohol is greater in those with AUD compared to moderate drinkers, consistent with the concept of alcohol 'priming microglia'.
  Interventions: Drug: Oral Alcohol Challenge

INTERVENTIONS:
Drug: Oral Alcohol Challenge — Subjects will drink an alcohol dose designed to achieve a BAL of 0.08

SUMMARY:
This study uses positron emission tomography imaging of the 18-kDa translocator protein to measure the brain's immune response to alcohol.

DETAILED DESCRIPTION:
Alcohol Use Disorder affects nearly 14% of the population, accruing considerable cost to individual families and society. Much of this cost stems from alcohol's influence on the immune system. Alcohol impairs peripheral immune function, evidenced by increased susceptibility to infection related diseases such as liver cirrhosis and pancreatitis. The neuroimmune consequences of alcohol are subtler. Preclinically, alcohol triggers neuroimmune abnormalities that contribute to cognitive dysfunction, neurodegeneration, and alter alcohol drinking behaviors. Yet, limited experimental tools hamper translational efforts to study alcohol's effects on neuroimmune function in people. We propose to address this deficit by developing an innovative human imaging paradigm that measures neuroimmune response to alcohol.

ELIGIBILITY:
General Inclusion Criteria:

1. Men and women, aged 21-50 years
2. Willing and able to give voluntary written informed consent
3. Able to read and write English and communicate effectively with the investigators, and comply with all study requirements, restrictions, and directions of the clinic staff
4. AUD Subjects will meet DSM-5 criteria for current Alcohol Use Disorder
5. Moderate Drinkers will report consuming alcohol on at least one occasion in the past three months that would result in an estimated blood alcohol level greater than 100 mg/dl but not meet DSM-5 criteria for AUD. This is to ensure that subjects have prior drinking exposure consistent with levels proposed in this study. Prospective subjects will be asked to recall the heaviest two days of drinking in the previous three months. Using this information, approximate BAC will be calculated for those prior episodes.
6. Medically healthy upon physical examination and laboratory testing.

General Exclusion Criteria:

1. Individuals whom the investigators deem may not be able to comply with alcohol abstinence for 48 hours prior to study day.
2. Current significant medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology.
3. History of or current neurological or significant psychiatric disorder such as schizophrenia or bipolar disorder (DSM-5 Axis 1).
4. Other substance use disorder with the exception of nicotine dependence in smokers as assessed with the SCID or positive urine screen for drugs of abuse.
5. Participants with any significant current medical conditions that would contraindicate the consumption of alcohol, such as history of neurological trauma or diseases, seizures, delirium or hallucinations, hepatic, or other unstable medical conditions.
6. Current suicidal or homicidal intent or behavior, or history of suicidal or homicidal behavior.
7. No barbiturates or other known microsomal enzyme induces or inhibitors in the past month.
8. History of significant head trauma.
9. Women who are pregnant or nursing or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD).
10. Regular or current significant use of any prescription, herbal or illegal psychotropic medications (e.g., antidepressants, antipsychotics, anxiolytics, ecstasy) in the past 6 mo, with no current illegal drug use confirmed by urine toxicology (except for cocaine and marijuana when relevant).
11. Have MRI-incompatible implants and other contraindications for MRI, such as a pacemaker, artificial joints, non-removable body piercings, claustrophobia, etc.
12. Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
13. Subjects with current, past or anticipated exposure to radiation in the work place within one year of proposed research PET scans.
14. Subjects with history of IV drug use which would prevent venous access for PET tracer injection.
15. Blood donation within eight weeks of the start of the study
16. History of blooding disorder or currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ansel T Hillmer, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Drinkers: Aim 1:
  A baseline PET scan with [11C]PBR28, a TSPO-specific radioligand, will be conducted with moderate drinkers. Next, subjects will drink a fixed alcohol dose, followed a post-alcohol [11C]PBR28 PET scan timed to capture acute neuroimmune response. [11C]PBR28 distribution volumes (VT), which are proportional to TSPO number, will be measured throughout the brain. We will test the hypothesis that acute alcohol robustly increases [11C]PBR28 VT, consistent with microglial activation. The percent change in [11C]PBR28 VT (ΔVT) from baseline will quantify the magnitude of neuroimmune response.
  Oral Alcohol Challenge: Subjects will drink an alcohol dose designed to achieve a BAL of 0.08
- Alcohol Use Disorder (AUD): Aim 2:
  AUD subjects will participate in the study design described in Aim 1 (a baseline [11C]PBR28 PET scan, drink a fixed alcohol dose, followed by a post-alcohol [11C]PBR28 PET scans). The magnitude of neuroimmune response, quantified by ΔVT, will be compared between moderate drinkers and individuals with AUD to test the hypothesis that the neuroimmune response to alcohol is greater in those with AUD compared to moderate drinkers, consistent with the concept of alcohol 'priming microglia'.
  Oral Alcohol Challenge: Subjects will drink an alcohol dose designed to achieve a BAL of 0.08
Period: Overall Study
Arm/Group | Moderate Drinkers | Alcohol Use Disorder (AUD)
Started | 11 | 3
Completed | 9 | 3
Not Completed | 2 | 0
Not completed — Arterial Line Failure, unable to proceed with PET scan | 2 | 0

BASELINE CHARACTERISTICS:
Population: Moderate Drinkers will self-report drinking consistent with at least one binge alcohol event in the past three months but will not meet DSM-5 criteria for AUD to ensure that accustomed drinking levels are not exceeded in the laboratory. AUD subjects will meet DSM-5 criteria for current Alcohol Use Disorder.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Drinkers | Alcohol Use Disorder (AUD) | Total
Number analyzed (Participants) | 11 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.36 (7.84) | 34.33 (7.76) | 31.21 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
rs6971 Genotype [Count of Participants; unit: Participants] — This rs6971 genotype is a well-characterized polymorphism that directly affects the radiotracer affinity for the TSPO site. Study participants are prospectively genotyped. Low Affinity Binders (LAB, homozygotes for the minor allele, ~10% of the population) are excluded due to limited image quality. MAB or HAB status is included as a fixed factor in final statistical analyses.
  Participants
    High Affinity Binder (HAB) | 10 | 1 | 11
    Mixed Affinity Binder (MAB) | 1 | 2 | 3
    Low Affinity Binder (LAB) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in [11C]PBR28 Distribution Volume After Alcohol Challenge.
Description: This is the percent change in [11C]PBR28 distribution volume (V_T) post-alcohol relative to baseline.
  This is calculated as [V_T(Post-Alcohol) - V_T(Baseline)]/V_T(Baseline)
  As a percent change, it could range from -10% to 200%.
Time Frame: The post-alcohol imaging scan start will begin between one and fours hours after the oral alcohol challenge is completed. The total scan time for each imaging scan is 120 minutes long.
Population: The ten participants (7M, 3F; 3 Mild AUD) who completed the laboratory drinking session were included in whole-body PET and cytokine data analysis.
Measure: Mean (Standard Deviation); unit: [11C]PBR28 VT (% change)
Arm/Group | Moderate Drinkers | Alcohol Use Disorder (AUD)
Number analyzed (Participants) | 7 | 3
[11C]PBR28 VT (% change) | 15.79 (8.00) | 6.36 (1.27)

ADVERSE EVENTS:
Time Frame: 1 Month After Study Day
Arm/Group | Moderate Drinkers | Alcohol Use Disorder (AUD)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 0/11 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04251221/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04251221/ICF_001.pdf